CLINICAL TRIAL: NCT05301101
Title: High Dose Re-Irradiation Utilizing Advanced Deformable Image Registration (DIR) and Individualized Organ At Risk (OAR) Dose Calculations With Organ Specific Toxicity Analysis (REDIRICT)
Brief Title: High Dose Re-Irradiation Utilizing Advanced Deformable Image Registration (DIR) and Individualized Organ At Risk (OAR) Dose Calculations With Organ Specific Toxicity Analysis
Acronym: REDIRICT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Elizabeth Gore, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00042951
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
Keywords: high dose radiation; re-irradiation
MeSH Terms: interventions — Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cancer patients receiving definitive radiation therapy with overlap of a previously treated field (Experimental): This is a re-irradiation study in solid tumor patients receiving definitive high dose radiation therapy to treatment volumes that include overlap with previously irradiated organs at risk.
  Interventions: Radiation: Re-irradiation

INTERVENTIONS:
Radiation: Re-irradiation — Patients will undergo re-irradiation following treatment planning based on current standard practice as determined by treating physicians and multidisciplinary teams.

SUMMARY:
This trial applies a uniform approach to re-irradiation for planning and diagnostic image fusion, dose summation, dose calculations, and follow up for tumor control and detailed toxicity analysis of serial Organs At Risk (OARs). Serial organs include named arteries and nerves, spinal cord, and gastrointestinal tract.

DETAILED DESCRIPTION:
STUDY DESIGN: For each serial OAR, we expect that 10% or less of reirradiated patients will have a Grade 3-5 toxicity. Under this assumption, 15 patients treated at a defined OAR will provide a 90% confidence interval (CI) for the Grade 3-5 OAR toxicity rate with a CI width no larger than 29%. A total of 120 treated patients (15 per OAR) are needed to provide this level of precision for toxicity rates within all 8 OARs (spinal cord, brachial plexus, named vessels, esophagus, duodenum, rectum, proximal bronchus/trachea, liver).

For each OAR, the numbers of patients reirradiated and Grade 3-5 toxicities among them will be tabulated. The Grade 3-5 toxicity rate among treated patients will be estimated separately for each OAR using the sample proportion and a 90% Wilson score confidence interval. Only patients who initiate re-irradiation therapy will be included in this analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent
2. Patients ≥18 years of age receiving definitive or postoperative high dose radiation to volume that includes overlap with previously irradiated OAR(s).
3. Prior radiation dosimetry must be available.
4. Participants must have stage I-IV biopsy proven solid malignancy (histologic proof or unequivocal cytologic proof solid tumor malignancy from either the primary or any metastatic site). Documentation of pathology reports are required. Local review of pathology or cytology is at the discretion of the multidisciplinary team.
5. Histologic confirmation of target lesion recurrence is recommended.
6. Documentation of consensus for recommendation of reirradiation by multidisciplinary team and location of target lesion or postoperative site to be treated.
7. Documentation of whether or not concurrent cancer therapy drugs are recommended and rationale.
8. Documentation of rationale for not obtaining tissue confirmation of the target lesion, if applicable.
9. Baseline target lesion imaging with CT, positron emission tomography (PET) /CT, or MRI is required within six weeks of trial enrollment. CT or MRI simulation scans may be used for baseline imaging.
10. Patients who have had disease resected in a previously irradiated field and are at high pathological and clinical risk for recurrence as defined by the treating Radiation Oncologist and multidisciplinary team, are eligible for study.
11. Measurable disease is not required for patients being treated postoperatively.
12. Baseline labs are per standard practice. Values will be dependent on the OARs being treated. (Per standard practice, radiation therapy volumes to OARs are modified to accommodate compromised renal, liver, pulmonary or other OAR function). Recommended labs and values include:

    * Aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 x upper limit of normal (ULN) or < 5 x ULN with metastatic liver disease.
    * Total bilirubin < 1.5 x ULN
    * Absolute neutrophil count (ANC) > 500 cells/mm^3
    * Platelets > 50,000 cells/mm^3
    * Creatinine < 1.5 x ULN or Creatinine clearance > 45 mL/min if creatinine is > 1.5 x ULN (calculated Creatinine Clearance (CrCl) based on Cockcroft-Gault equation)
13. Eastern Cooperative Oncology Group (ECOG) Performance Score 0-2.
14. Patients must have resolution of acute toxic effect(s) of most recent cancer therapy to Grade 1 or 2.
15. Life expectancy of at least 6 months.
16. Female patients of childbearing potential must have negative urine or serum pregnancy test within 7 days prior to start of re-irradiation.
17. Ability to complete the self-reported questionnaires (translations will be made available if the patient's primary language is not English).
18. Concurrent participation on pharmaceutical, investigator-initiated, National Clinical Trials Network (NCTN), or other multisite clinical trials that include re-irradiation is allowed.

Exclusion Criteria:

1. Patients receiving low dose radiation for symptom management only.
2. Patients with evidence of severe or uncontrolled systemic conditions.
3. Life expectancy of less than 6 months.
4. ECOG Performance status ≥ 3.
5. Women of childbearing potential who are known to be pregnant or are unwilling to use an acceptable method of contraception from the time of informed consent until completion of the course of radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Organ-specific grade 3 toxicity. | Up to 24 months
  The number of patients with organ-specific grade 3 toxicity in patients undergoing high-dose re-irradiation. Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 will be used to define the grade.
Organ-specific grade 4 toxicity. | Up to 24 months
  The number of patients with organ-specific grade 4 toxicity in patients undergoing high-dose re-irradiation. Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 will be used to define the grade.
Organ-specific grade 5 toxicity. | Up to 24 months
  The number of patients with organ-specific grade 5 toxicity in patients undergoing high-dose re-irradiation. Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 will be used to define the grade.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gore, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No